CLINICAL TRIAL: NCT01436253
Title: Non-Interventional Study In Hyperlipidemic Patients Who Do Not Reach Satisfactory Lipid Values With Existing Hypolipemic Therapy
Brief Title: Study of Lipid Control in Hyperlipidemic Participants (MK-0653-179)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0653-179
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Croatian participants with hyperlipidemia: Participants being treated in a physician's office for hyperlipidemia who have not achieved target lipid levels on their current hypolipemic therapy.
  Interventions: Behavioral: Lifestyle Changes; Drug: Hypolipemics

INTERVENTIONS:
Behavioral: Lifestyle Changes — Diet, increased physical activity, and weight reduction as per European Guidelines on the Management of Hypercholesterolemia accepted by the Croatian Society of Cardiology were encouraged in addition to pharmacological measures at the discretion of the treating physician.
Drug: Hypolipemics — Pharmacological measures at the discretion of the treating physician and in accordance with the respective authorized label and European Guidelines on the Management of Hypercholesterolemia accepted by the Croatian Society of Cardiology.

SUMMARY:
This study is being done to see whether dietary and medicinal measures compliant with hyperlipidemia treatment guidelines will result in achieving target lipid values and to evaluate the total risk of cardiovascular disease in study participants who have not reached satisfactory lipid levels with their current hypolipemic therapy.

ELIGIBILITY:
Inclusion criteria:

* Hyperlipidemic
* On therapy for hyperlipidemia for >=3 months without achieving target lipid values

Exclusion criteria:

* Hypersensitivity or intolerance to hypolipemics
* Significant myopathy or rhabdomiolysis probably caused by hypolipemics
* Uncontrolled endocrine or metabolic disease which is known to affect lipid or lipoprotein values (for example, hypothyroidism and hyperthyroidism)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Croatian participants with inadequately controlled hyperlipidemia being treated in the primary care setting
Sampling Method: Non-Probability Sample
Enrollment: 2196 (Actual)
Dates: Start 2008-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants in Croatia being treated in Physician Offices for hyperlipidemia who have not achieved target lipid levels on their current therapy.
Period: Overall Study
Arm/Group | All Participants
Started | 2196
Completed | 1897
Not Completed | 299
Not completed — Lost to Follow-up | 182
Not completed — Not meeting all eligibility criteria | 117

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 1897
Age, Customized [Number; unit: Participants] — Participants meeting all inclusion and exclusion criteria.
  Participants
    30-44 Years | 118
    45-64 Years | 1063
    >=65 Years | 716
Sex/Gender, Customized [Number; unit: Participants] — Participants meeting all inclusion and exclusion criteria.
  Participants
    Female | 1042
    Male | 770
    Unknown | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Target Lipid Values
Description: Target total cholesterol value was <4.5 mmol/L and target low densisty lipoprotein (LDL) value was <2.5 mmol/L
Time Frame: Baseline and Month 3
Population: Participants meeting all inclusion and exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: Participants in Croatia being treated in Physician Offices for hyperlipidemia who have not achieved target lipid values on their current therapy.
Arm/Group | All Participants
Number analyzed (Participants) | 1897
Percentage of participants | 46.8 [44.6 to 49.0]

2. Primary Outcome: Percentage of Participants With Reduced Cardiovascular Risk
Description: Cardiovascular risk assessment to determine the 10-year risk for developing cardiovascular disease was done using Framingham risk scoring; categories scored are age, high density lipoprotein (HDL) cholesterol value, total cholesterol value, history of cigarette smoking, and systolic blood pressure. The total of all the points for each risk factor is used to assign a percentage of risk for the occurence of cardiovascular disease within 10 years. Total points for men range from -9 to +37 and for women from -8 to +46; >=17 total points for men, and >=25 total points for women indicates a >=30% risk of developing cardiovascular disease.
Time Frame: Baseline and Month 3
Population: Participants meeting all inclusion and exclusion criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 1897
Percentage of participants | 51.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 3 months, starting with the first visit and ending with the final visit to the Physician's office.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/2196
Other Adverse Events (participants affected / at risk) | 0/2196

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No Investigator may publish or disclose any study information without permission from the Sponsor.